CLINICAL TRIAL: NCT03518684
Title: Obstetrical Gel Use to Shorten Labor and Prevent Lower Genital Tract Trauma: A Randomized Controlled Trial
Brief Title: Obstetrical Gel Use to Shorten Labor and Prevent Lower Genital Tract Trauma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Elie Hobeika, Assistant Professor of Clinical Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OGY.EH.03
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Labor Stage, Second
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: In this randomized controlled study, the patients will be randomly assigned to either Group 1 in which they will receive the standard care during labor and delivery without the use of the obstetrical gel or Group 2 in which they will have the standard care during labor and delivery with the vaginal application of the obstetrical gel according to the study protocol. Those 2 groups will be further divided into 4 subgroups where the parity will be accounted for (nulliparous [never delivered beyond 20 weeks of gestation in a previous pregnancy] or primiparous or more). Based on our departmental statistics, ~90% of laboring patients receive epidural. Hence receiving an epidural will not have a major impact on the duration of the second stage of labor; yet, whether the patient received epidural or not will be adjusted for.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (No Intervention): Group 1 in which they will receive the standard care during labor and delivery without the use of the obstetrical gel
- Group 2 (Experimental): Group 2 in which they will have the standard care during labor and delivery with the vaginal application of the obstetrical gel according to the study protocol. Those 2 groups will be further divided into 4 subgroups where the parity will be accounted for (nulliparous [never delivered beyond 20 weeks of gestation in a previous pregnancy] or primiparous or more)
  Interventions: Drug: Natalis

INTERVENTIONS:
Drug: Natalis — A specially-designed sterile obstetric gel (Natalis) will be used for this trial. The obstetric gel is a birth gel with no pharmacologic effects that has a purely physical activity. It contains propylene glycol, glycerol, sodium chloride, xanthan gum, hydroxyethylcellulose and water.
  Starting with the first vaginal examination the obstetric gel will be used. After each vaginal examination, 3-5 mL of obstetric gel will be introduced into the vaginal birth canal in the area in front of the child using the sterile obstetric gel applicator without any manipulation or massaging. Additional obstetric gel will be added 15-30 minutes after rupture of the membranesOnce the head of the child is visible, the mouth and nose region will be wiped clean. A dry towel will be used to liberate the child in order to prevent the child from slipping
  Arms: Group 2

SUMMARY:
Recent literature shows that birth injury is associated with postpartum pelvic floor dysfunction (pelvic organ prolapse and fecal and urinary incontinence). Prolonged labor, namely during the 2nd stage, is one of the main obstetric risk factors responsible for anal sphincter rupture and fecal incontinence. In addition, it is associated with increased maternal and neonatal morbidities including increased risk of lower genital tract lacerations. In an effort to shorten labor and decrease lower genital tract trauma many techniques have been investigated.

The objective of our study is to investigate whether the use of obstetric gel shortens the first and second stage of labor and exerts a protective effect on the lower genital tract. Neonatal and maternal morbidities will be also assessed.

The study design will be a randomized controlled trial of 2 groups, where the patients presenting for vaginal delivery will be randomly assigned to either:

* Group 1 who will receive the standard care during labor and delivery
* Group 2 who will receive the standard care during labor and delivery with the vaginal application of the obstetrical gel The goal of this randomized controlled study is to compare the length of the first and 2nd stage of labor and the lower genital tract integrity in the 2 groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Intended vaginal delivery
* Singleton baby in vertex presentation
* Low risk pregnancy at term (37-42 weeks of gestation)
* Estimated birth weight between 2000 g and 4500 g (clinically or by sonography)
* Signed written informed consent

Exclusion Criteria:

* Contraindications for vaginal delivery (placenta previa, active herpes infection, etc…)
* Advanced cervical dilation (≥ 5 cm)
* Suspected amniotic infection (fever, foul smelling discharge, fetal tachycardia, abdominal pain)
* Non reassuring fetal heart tracing
* Prolonged rupture of the membranes (24 hours)
* Suspected major fetal malformations
* Suspected cephalopelvic disproportion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in the length of the second stage of labor | Second stage of labor, a reduction to 39.9 minutes from a calculated average of 66.5 minutes
  40% reduction in the duration of the second stage of labor with a calculated average duration of 66.5 min. Thus a reduction to 39.9 minutes for every patient recruited

CONTACTS AND LOCATIONS:
Locations (1):
- Amercian University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR